CLINICAL TRIAL: NCT06082414
Title: Systemic Management in Extremely Preterm and Extremely Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other); Peking University Third Hospital (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); Peking Union Medical College Hospital (Other); Beijing Children's Hospital (Other); Beijing Friendship Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); The Second Hospital of Hebei Medical University (Other); Handan Central Hospital (Other); Xingtai People's Hospital (Other); Tianjin Medical University General Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Children's Hospital of Hebei Province (Other); Tianjin First Central Hospital (Other); Chifeng Municipal Hospital (Other); Tianjin Medical University Second Hospital (Other); PLA Rocket Force Characteristic Medical Center (Other)
Responsible Party: Principal Investigator, Li Shuaijun, Post doctor, Attending physician, Peking University
Other Study IDs: 2019(21)
Record Dates: First submitted 2023-10-04; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Bronchopulmonary Dysplasia; Death
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- <28 weeks and <1000 grams: By gestational age and birth weight, infants were classified into 3 groups. No interventions because of an observational study.
  Interventions: Other: no interventions
- <28 weeks and ≥1000 grams: By gestational age and birth weight, infants were classified into 3 groups. No interventions because of an observational study.
  Interventions: Other: no interventions
- ≥28 weeks and <1000 grams: By gestational age and birth weight, infants were classified into 3 groups. No interventions because of an observational study.
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions because of an observational study

SUMMARY:
to estimate incidences of major complications, such as bronchopulmonary dysplasia, death, and delivery room resuscitation among extremely preterm and extremely low birth weight infants in Northern China

DETAILED DESCRIPTION:
to estimate incidences and risk factors of bronchopulmonary dysplasia, death, and delivery room resuscitation among extremely preterm and extremely low birth weight infants in Northern China

ELIGIBILITY:
Inclusion Criteria:

1. born between January 1, 2015, and December 31, 2018;
2. a birth weight <1000grams or a gestational age <28 weeks;
3. admitted within 72 hours after birth.

Exclusion Criteria:

No medical history in the electronic record

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants with a birth weight <1000grams or a gestational age <28 weeks;
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
incidences | at 36 weeks' corrected age (CA) or at discharge
  to investigate incidences of bronchopulmonary dysplasia
risk factors | at 36 weeks' corrected age (CA) or at discharge
  to investigate risk factors of bronchopulmonary dysplasia
incidences of delivery room resuscitation | on admission
  to investigate incidences of delivery room resuscitation
risk factors of delivery room resuscitation | on admission
  to investigate risk factors of delivery room resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Qi Feng, Study Chair — Peking University First Hospital
Locations (1):
- Qi Feng, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li S, Feng Q, Huang X, Tian X, Zhou Y, Ji Y, Zhai S, Guo W, Zheng R, Wang H. Association of different doses of antenatal corticosteroids exposure with early major outcomes and early weight loss percentage in extremely preterm infants or extremely low birthweight infants: a multicentre cohort study. BMJ Paediatr Open. 2024 Jun 18;8(1):e002506. doi: 10.1136/bmjpo-2024-002506. PMID 38897621